CLINICAL TRIAL: NCT05261230
Title: Trauma Focused Vedic Counselling for Women Victims of Domestic Abuse: Community-based Pilot Study.
Brief Title: Vedic Counselling for Women Victims of Domestic Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Active Natural Limited (Industry)
Collaborators: NMP Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANL/GS/001
Record Dates: First submitted 2022-02-19; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Intimate Partner Violence; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vedic Counselling Group (Experimental): Vedic Counselling was given by trained and experienced therapists
  Interventions: Behavioral: Vedic Counselling
- Usual Care Group (Active Comparator): Standard psychosocial care delivered by psychologists.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Vedic Counselling — Trauma focused Vedic Counselling intervention was delivered by trained and experienced therapist of Yoga and Vedanta.12-week sessions were provided on one to one bases on personalised approach.
  Arms: Vedic Counselling Group
Behavioral: Standard Care — The active control group received standard psychosocial care provided by the participating psychologists and psychiatrists.
  Arms: Usual Care Group

SUMMARY:
The Vedic Counselling is the whole person approach, system of total life style counselling based on 'Vedic Laws of right living, right actions, right relationship and right awareness'.Vedic Counselling was developed as trauma focused therapy for this study to treat female victims of domestic abuse.

ELIGIBILITY:
Inclusion Criteria:

* Female survivors of Domestic Abuse
* 18 years old or older
* Sign informed consent

Exclusion Criteria:

* Severe mental illness that requires specialized treatment
* Terminally ill
* Under psychiatric medication
* Chronic illnesses

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 66 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Symptoms of Post-Traumatic Stress Disorders (PTSD) | Change from baseline PTSD symptoms at 12-weeks
  PTSD symptoms measured by revised version of the Impact of Event Scale (IES-r) 22 questions and a scoring range of 0 to 88

SECONDARY OUTCOMES:
Symptoms of Anxiety | Change from baseline anxiety at 12-weeks
  Anxiety was measured through Depression Anxiety Stress Scale (DASS)-21, self-report questionnaire consisting of 21 items, 7 items per subscale: scored 0 to 3 on each item.
Symptoms of Depression | Change from baseline depression at 12-weeks
  Depression was measured through Depression Anxiety Stress Scale (DASS)-21
Symptom of Stress | Change from baseline stress at 12-weeks
  Stress was measured through Depression Anxiety Stress Scale (DASS)-21
Self-Esteem | Change from baseline at 12 weeks
  Self-esteem was measured using the Rosenberg's Self-Esteem Scale. Each question response that gives a score between 1-4.

CONTACTS AND LOCATIONS:
Overall Officials: Sadhana Sharma, Principal Investigator — Gyansanjeevani
Locations (1):
- NMP Medical Research Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided